CLINICAL TRIAL: NCT04003103
Title: A Phase 2a, Double-Blind, Placebo-Controlled Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of Oral MK-8591 Once-Monthly in Participants at Low- Risk for HIV-1 Infection
Brief Title: Safety and Pharmacokinetics of Oral Islatravir (MK-8591) Once Monthly in Participants at Low Risk of Human Immunodeficiency Virus 1 (HIV-1) Infection (MK-8591-016)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 8591-016; Merck Protocol Number (Other: MK-8591-016); 2019-001704-38 (EudraCT Number)
Record Dates: First submitted 2019-06-27; First posted 2019-07-01 (Actual); Results first posted 2023-03-21 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: HIV-1 Infection
MeSH Terms: interventions — islatravir

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Islatravir 60 mg (Experimental): 60 mg islatravir + placebo for islatravir administered once monthly, orally in capsule form for 24 weeks
  Interventions: Drug: Islatravir; Drug: Placebo
- Islatravir 120 mg (Experimental): 120 mg islatravir administered once monthly, orally in capsule form for 24 weeks
  Interventions: Drug: Islatravir
- Placebo (Placebo Comparator): Placebo for islatravir administered once monthly, orally in capsule form for 24 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Islatravir — Islatravir 30 mg capsules taken by mouth.
  Other Names: MK-8591
  Arms: Islatravir 120 mg; Islatravir 60 mg
Drug: Placebo — Placebo capsules taken by mouth.
  Arms: Islatravir 60 mg; Placebo

SUMMARY:
This study will evaluate the safety, tolerability and pharmacokinetics (PK) of 6 once-monthly doses of oral islatravir (60 mg and 120 mg) compared with placebo in adults at low risk of HIV-1 infection

DETAILED DESCRIPTION:
This study is ongoing for collection of safety follow-up of infants born to mothers participating in the study. The present results are based on the Week 68 interim analysis.

ELIGIBILITY:
Inclusion Criteria:

* Is in general good health with acceptable laboratory values at screening
* Is confirmed HIV-uninfected based on negative HIV-1/HIV-2 test result before randomization
* Has low risk of HIV infection, within 12 months prior to screening visit or the rescreening visit (if applicable)
* Use contraceptives consistent with local regulations
* Female is not pregnant or breastfeeding, and is not a woman of childbearing potential (WOCBP)
* A WOCBP is using an acceptable contraceptive method, or is abstinent from heterosexual intercourse as their preferred and usual lifestyle; or has a negative pregnancy test.

Exclusion Criteria:

* Has hypersensitivity or other contraindication to any of the components of the study interventions as determined by the investigator
* Has an active diagnosis of hepatitis due to any cause
* Has a history of malignancy ≤5 years prior to signing informed consent except for adequately treated basal cell or squamous cell skin cancer or in situ cervical cancer.
* Is taking or is anticipated to require systemic immunosuppressive therapy, immune modulators, or any prohibited therapies from 30 days prior to Day

  1 through the duration of the study.
* Is currently participating in or has participated in an interventional clinical study with an investigational compound or device within 30 days prior to Day1 through the duration of the study.
* Has previously been randomized in a study and received islatravir (MK-8591).
* Female is expecting to conceive or donate eggs at any time during the study
* Has QTc interval (using Fridericia correction) >450 msec (for males) or >460 msec (for females) or deemed clinically abnormal by the investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 242 (Actual)
Dates: Start 2019-09-19 (Actual); Primary Completion 2022-03-18 (Actual); Study Completion 2022-11-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (9):
- United States (4):
  - Research Centers of America, LLC ( Site 0007), Hollywood, Florida
  - Johns Hopkins School of Medicine - Drug Development Unit ( Site 0002), Baltimore, Maryland
  - Celerion, Inc. ( Site 0006), Lincoln, Nebraska
  - Magee Womens Research Institute ( Site 0001), Pittsburgh, Pennsylvania
- Israel (2):
  - Hadassah Ein Karem Jerusalem ( Site 0016), Jerusalem, Jerusalem
  - Rambam Medical Center ( Site 0017), Haifa
- South Africa (3):
  - JOSHA Research ( Site 0015), Bloemfontein, Free State
  - Clinical HIV Research Unit CHRU ( Site 0014), Johannesburg, Gauteng
  - Emavundleni Vaccine Centre ( Site 0011), Cape Town, Western Cape

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- [Result] Hillier SL, Bekker LG, Riddler SA, Hendrix CW, Badal-Faesen S, Macdonald P, Nair G, Lombaard J, Caraco Y, Peer A, Patel M, Vargo R, Homony B, Nedrow K, Evans B, Wickremasingha P, Zhou YP, Teal V, Hwang P, McMullan C, Kaufman KD, Robertson MN, Plank RM. Safety, Tolerability, and Pharmacokinetics of Once-Monthly Oral Islatravir: A Phase 2a Study in Participants at Low Risk for Acquiring Human Immunodeficiency Virus Type 1. J Infect Dis. 2025 Nov 14;232(5):1050-1060. doi: 10.1093/infdis/jiaf222. PMID 40327547
- [Derived] Pham M, Wickremasingha P, Vargo R, Patel M, Nedrow K, Homony B, Robertson MN, Plank RM. Brief Report: Exploratory Substudy of a Phase 2 Trial to Evaluate the Pharmacokinetic Effect of Once-Monthly Islatravir on Long-Acting Reversible Contraceptives. J Acquir Immune Defic Syndr. 2025 Aug 1;99(4):374-378. doi: 10.1097/QAI.0000000000003678. PMID 40260892
- [Derived] Devanathan AS, Cottrell ML. Pharmacology of HIV Cure: Site of Action. Clin Pharmacol Ther. 2021 Apr;109(4):841-855. doi: 10.1002/cpt.2187. Epub 2021 Mar 5. PMID 33540481
- See also: Merck Clinical Trials Information — http://www.merckclinicaltrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Healthy HIV-uninfected male and female participants were enrolled at 9 study centers in 3 countries.
Groups:
- Islatravir 60 mg: Participants receive two ISL 30 mg capsules + two ISL placebo capsules once monthly from Day 1 to Week 24 plus 12 weeks of follow-up in the Treatment Phase. The Extended Follow-up Phase is from Week 36 to Week 68.
- Islatravir 120 mg: Participants receive four ISL 30 mg capsules once monthly from Day 1 to Week 24 plus 12 weeks of follow-up in the Treatment Phase. The Extended Follow-up Phase is from Week 36 to Week 68.
- Placebo: Participants receive four placebo capsules once monthly from Day 1 to Week 24 plus 12 weeks of follow-up in the Treatment Phase. The Extended Follow-up Phase is from Week 36 to Week 68.
Period: Overall Study
Arm/Group | Islatravir 60 mg | Islatravir 120 mg | Placebo
Started | 97 | 97 | 48
Completed | 82 | 91 | 45
Not Completed | 15 | 6 | 3
Not completed — Death | 1 | 0 | 0
Not completed — Lost to Follow-up | 4 | 3 | 2
Not completed — Withdrawal by Subject | 10 | 1 | 1
Not completed — Status not recorded | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Islatravir 60 mg | Islatravir 120 mg | Placebo | Total
Number analyzed (Participants) | 97 | 97 | 48 | 242
Age, Continuous [Mean (Standard Deviation); unit: Years] | 33.6 (9.9) | 33.2 (9.7) | 30.9 (7.9) | 32.9 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 66 | 64 | 33 | 163
  Male | 31 | 33 | 15 | 79
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 19 | 9 | 8 | 36
  Not Hispanic or Latino | 78 | 88 | 40 | 206
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 1
  Asian | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 37 | 48 | 16 | 101
  White | 55 | 44 | 29 | 128
  More than one race | 5 | 3 | 3 | 11
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With ≥1 Adverse Event (AE) Through Week 36
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
Time Frame: Up to 36 weeks
Population: All participants who received ≥1 dose of study therapy are included.
Measure: Count of Participants; unit: Participants
Arm/Group | Islatravir 60 mg | Islatravir 120 mg | Placebo
Number analyzed (Participants) | 97 | 97 | 48
Participants | 66 | 63 | 36

2. Primary Outcome: Number of Participants Discontinuing From Study Therapy Due to AE
Description: as for outcome 1
Time Frame: Up to 20 weeks
Population: All participants who received ≥1 dose of study therapy are included.
Measure: Count of Participants; unit: Participants
Arm/Group | Islatravir 60 mg | Islatravir 120 mg | Placebo
Number analyzed (Participants) | 97 | 97 | 48
Participants | 1 | 1 | 0

3. Primary Outcome: Number of Participants Discontinuing From Study Therapy Due to ≥1 Drug-related AE
Description: A drug-related AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, that is considered related to the study therapy.
Time Frame: Up to 20 weeks
Population: All participants who received ≥1 dose of study therapy are included.
Measure: Count of Participants; unit: Participants
Arm/Group | Islatravir 60 mg | Islatravir 120 mg | Placebo
Number analyzed (Participants) | 97 | 97 | 48
Participants | 1 | 1 | 0

4. Primary Outcome: Number of Participants With ≥1 Drug-related AE Through Week 36
Description: A drug-related AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, that is considered related to the study intervention.
Time Frame: Up to 36 weeks
Population: All participants who received ≥1 dose of study therapy are included.
Measure: Count of Participants; unit: Participants
Arm/Group | Islatravir 60 mg | Islatravir 120 mg | Placebo
Number analyzed (Participants) | 97 | 97 | 48
Participants | 9 | 14 | 12

5. Primary Outcome: Number of Participants With ≥1 Serious Adverse Event (SAE) Through Week 36
Description: An SAE is defined as any untoward medical occurrence that, at any dose, results in death; is life-threatening; requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent or significant disability/incapacity; is a congenital anomaly/birth defect; or is an other important medical event.
Time Frame: Up to 36 weeks
Population: All participants who received ≥1 dose of study therapy are included.
Measure: Count of Participants; unit: Participants
Arm/Group | Islatravir 60 mg | Islatravir 120 mg | Placebo
Number analyzed (Participants) | 97 | 97 | 48
Participants | 1 | 0 | 0

6. Primary Outcome: Number of Participants With a ≥1 Grade 3 to Grade 5 AE up to Week 36
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study therapy, whether or not considered related to the study intervention. Toxicity grading was according to the National Institutes of Health Division of AIDS (NIH DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events version 2.1 (Grade 3 is 'severe'; Grade 4 is 'potentially life-threatening'; and Grade 5 'results in death').
Time Frame: Up to 36 weeks
Population: All participants who received ≥1 dose of study therapy are included.
Measure: Count of Participants; unit: Participants
Arm/Group | Islatravir 60 mg | Islatravir 120 mg | Placebo
Number analyzed (Participants) | 97 | 97 | 48
Participants | 5 | 4 | 1

7. Primary Outcome: Number of Participants With ≥1 Drug-related SAE Through Week 36
Description: An drug-related SAE is defined as any untoward medical occurrence that, at any dose, results in death; is life-threatening; requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent or significant disability/incapacity; is a congenital anomaly/birth defect; or is an other important medical event, that is considered related to study therapy.
Time Frame: Up to 36 weeks
Population: All participants who received ≥1 dose of study therapy are included.
Measure: Count of Participants; unit: Participants
Arm/Group | Islatravir 60 mg | Islatravir 120 mg | Placebo
Number analyzed (Participants) | 97 | 97 | 48
Participants | 0 | 0 | 0

8. Primary Outcome: Number of Participants With ≥1 Drug-related Grade 3 to 5 AE Through Week 36
Description: A drug-related Grade 3 to Grade 5 AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention; has a toxicity Grade 3 (severe), 4 (potentially life-threatening), or 5 (results in death); and is considered related to study therapy. Toxicity grading was according to the NIH DAIDS Table for Grading the Severity of Adult and Pediatric Adverse Events (v. 2.1).
Time Frame: Up to 36 weeks
Population: All participants who received ≥1 dose of study therapy are included.
Measure: Count of Participants; unit: Participants
Arm/Group | Islatravir 60 mg | Islatravir 120 mg | Placebo
Number analyzed (Participants) | 97 | 97 | 48
Participants | 0 | 0 | 0

9. Primary Outcome: Number of Participants With an AE Resulting in Death Through Week 36
Description: as for outcome 1
Time Frame: Up to 36 weeks
Population: All participants who received ≥1 dose of study therapy are included.
Measure: Count of Participants; unit: Participants
Arm/Group | Islatravir 60 mg | Islatravir 120 mg | Placebo
Number analyzed (Participants) | 97 | 97 | 48
Participants | 0 | 0 | 0

10. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Dosing to 672 Hours Postdose (AUC0-672) of Plasma ISL
Description: The AUC0-672 of ISL after dosing on Day 1 and Day 140 is reported. Only ISL-treated participants are included in the PK analysis.
Time Frame: Day 1 and Day 140: predose and 30-min postdose. On Day 2 collect ~24 hours after Day 1 dose. On Weeks 4, 8, 12 and 16, collect predose. Weeks 1, 2, 3, 21, 22, 23 and 24: collect at any time during the study visit.
Population: ISL-treated participants with data available who complied with the protocol sufficiently to ensure that generated data are likely to exhibit the effects of treatment, according to the underlying scientific model, are included.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*umol/L
Arm/Group | Islatravir 60 mg | Islatravir 120 mg | Placebo
Number analyzed (Participants) | 93 | 96 | 0
hr*umol/L
  Day 1 | 7.88 (56.8) | 16.6 (50.5) |
  Day 140: number analyzed (Participants) | 82 | 92 | 0
  Day 140 | 21.2 (140.3) | 37.6 (136.6) |

11. Secondary Outcome: Maximum Plasma Concentration (Cmax) of ISL
Description: The Cmax of ISL after dosing on Day 1 and Day 140 is reported. Only ISL-treated participants are included in the PK analysis.
Time Frame: Day 1 and Week 20, collect predose and 30-min postdose. On Day 2 collect ~24 hours after Day 1 dose. On Weeks 4, 8, 12 and 16, collect predose. Weeks 1, 2, 3, 21, 22, 23 and 24: collect at any time during the study visit.
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µmol/L
Arm/Group | Islatravir 60 mg | Islatravir 120 mg | Placebo
Number analyzed (Participants) | 97 | 97 | 0
µmol/L
  Day 1 | 0.387 (279.9) | 0.954 (186.2) |
  Day 140: number analyzed (Participants) | 85 | 92 | 0
  Day 140 | 0.376 (597.7) | 0.792 (349.6) |

12. Secondary Outcome: Trough Plasma Concentration (Ctrough) of ISL
Description: The plasma Ctrough of ISL after dosing on Day 1 and Day 140 is reported. Only ISL-treated participants are included in the PK analysis.
Time Frame: Day 1 and Week 20: predose and 30-min postdose. Day 2: 24 hours post Day 1 dose. Weeks 1, 2, 3, 21, 22, 23 and 24: any time during the study visit. Weeks 4, 8, 12 and 16: predose.
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µmol/L
Arm/Group | Islatravir 60 mg | Islatravir 120 mg | Placebo
Number analyzed (Participants) | 92 | 95 | 0
µmol/L
  Day 1 | 0.000556 (36.6) | 0.00101 (37.0) |
  Day 140: number analyzed (Participants) | 85 | 92 | 0
  Day 140 | 0.000809 (37.0) | 0.000124 (42.0) |

13. Secondary Outcome: Apparent Plasma Terminal Half-life (t1/2) of ISL
Description: The plasma t1/2 of ISL after dosing on Day 140 is reported. Only ISL-treated participants are included in the PK analysis.
Time Frame: as for outcome 11
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Islatravir 60 mg | Islatravir 120 mg | Placebo
Number analyzed (Participants) | 81 | 92 | 0
Hours
  Day 1 | NA (NA) — Insufficient data available on Day 1. | NA (NA) — Insufficient data available on Day 1. |
  Day 140 | 175 (16.2) | 177 (19.8) |

14. Secondary Outcome: Number of Participants With ≥1 AE Through Week 24
Description: as for outcome 1
Time Frame: Up to 24 weeks
Population: All participants who received ≥1 dose of study therapy are included.
Measure: Count of Participants; unit: Participants
Arm/Group | Islatravir 60 mg | Islatravir 120 mg | Placebo
Number analyzed (Participants) | 97 | 97 | 48
Participants | 58 | 60 | 32

15. Secondary Outcome: Number of Participants With ≥1 Drug-related AE Through Week 24
Description: as for outcome 4
Time Frame: Up to 24 weeks
Population: All participants who received ≥1 dose of study therapy are included.
Measure: Count of Participants; unit: Participants
Arm/Group | Islatravir 60 mg | Islatravir 120 mg | Placebo
Number analyzed (Participants) | 97 | 97 | 48
Participants | 9 | 14 | 12

16. Secondary Outcome: Number of Participants With ≥1 SAE Through Week 24
Description: as for outcome 5
Time Frame: Up to 24 weeks
Population: All participants who received ≥1 dose of study therapy are included.
Measure: Count of Participants; unit: Participants
Arm/Group | Islatravir 60 mg | Islatravir 120 mg | Placebo
Number analyzed (Participants) | 97 | 97 | 48
Participants | 1 | 0 | 0

17. Secondary Outcome: Number of Participants With a ≥1 Grade 3 to Grade 5 AE up to Week 24
Description: as for outcome 6
Time Frame: Up to 24 weeks
Population: All participants who received ≥1 dose of study therapy are included.
Measure: Count of Participants; unit: Participants
Arm/Group | Islatravir 60 mg | Islatravir 120 mg | Placebo
Number analyzed (Participants) | 97 | 97 | 48
Participants | 3 | 3 | 1

18. Secondary Outcome: Number of Participants With ≥1 Drug-related SAE Through Week 24
Description: as for outcome 7
Time Frame: Up to 24 weeks
Population: All participants who received ≥1 dose of study therapy are included.
Measure: Count of Participants; unit: Participants
Arm/Group | Islatravir 60 mg | Islatravir 120 mg | Placebo
Number analyzed (Participants) | 97 | 97 | 48
Participants | 0 | 0 | 0

19. Secondary Outcome: Number of Participants With ≥1 Drug-related Grade 3 to 5 AE Through Week 24
Description: as for outcome 8
Time Frame: Up to 24 weeks
Population: All participants who received ≥1 dose of study therapy are included.
Measure: Count of Participants; unit: Participants
Arm/Group | Islatravir 60 mg | Islatravir 120 mg | Placebo
Number analyzed (Participants) | 97 | 97 | 48
Participants | 0 | 0 | 0

20. Secondary Outcome: Number of Participants With an AE Resulting in Death Through Week 24
Description: as for outcome 1
Time Frame: Up to 24 weeks
Population: All participants who received ≥1 dose of study therapy are included.
Measure: Count of Participants; unit: Participants
Arm/Group | Islatravir 60 mg | Islatravir 120 mg | Placebo
Number analyzed (Participants) | 97 | 97 | 48
Participants | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 36 weeks
Description: All treated participants are included.
Arm/Group | Islatravir 60 mg | Islatravir 120 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 1/97 | 0/97 | 0/48
Serious Adverse Events (participants affected / at risk) | 1/97 | 0/97 | 0/48
Other Adverse Events (participants affected / at risk) | 24/97 | 23/97 | 16/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Islatravir 60 mg (N=97) | Islatravir 120 mg (N=97) | Placebo (N=48)
Intentional self-injury (Psychiatric disorders) | 1 | 0 | 0
Loss of consciousness (Nervous system disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Islatravir 60 mg (N=97) | Islatravir 120 mg (N=97) | Placebo (N=48)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 3 (3) | 4 (4)
Diarrhoea (Gastrointestinal disorders) | 5 (5) | 4 (5) | 4 (4)
Nausea (Gastrointestinal disorders) | 5 (6) | 7 (7) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 4 (5) | 4 (4) | 3 (4)
Accidental overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 3 (3)
Alanine aminotransferase increased (Investigations) | 2 (3) | 0 (0) | 3 (3)
Blood pressure increased (Investigations) | 1 (2) | 5 (5) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 0 (0) | 3 (4)
Headache (Nervous system disorders) | 10 (27) | 9 (9) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If publication activity is not directed by the Sponsor, the investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission.

DOCUMENTS (2):
  • Study Protocol (2021-12-08): https://cdn.clinicaltrials.gov/large-docs/03/NCT04003103/Prot_000.pdf
  • Statistical Analysis Plan (2021-12-08): https://cdn.clinicaltrials.gov/large-docs/03/NCT04003103/SAP_001.pdf